CLINICAL TRIAL: NCT00799526
Title: Transplant of Epithelium Conjunctival Human Autologous Cultivated ex Vivo in Amniotic Membrane for the Treatment of Symblepharon
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Jose Alvaro Pereira Gomes, UNIFESP, SAO PAULO, SP, BRAZIL
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1075/08
Record Dates: First submitted 2008-11-28; First posted 2008-12-01 (Estimated); Last update posted 2008-12-01 (Estimated); Status verified 2008-11

CONDITIONS: Symblepharon
Keywords: Ex Vivo Conjunctival Epithelial Cell; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ex Vivo Transplantation (Experimental): Autologous Ex Vivo Conjunctival Epithelial Cell Expansion for Symblepharon Transplantation
  Interventions: Procedure: Autologous Ex Vivo Conjunctival for Symblepharon Transplantation; Procedure: Ex Vivo Conjunctival for Symblepharon Transplantation

INTERVENTIONS:
Procedure: Autologous Ex Vivo Conjunctival for Symblepharon Transplantation — Safety and efficacy of conjunctival ex vivo for reconstruction of the ocular surface.
Procedure: Ex Vivo Conjunctival for Symblepharon Transplantation — The safety and efficacy of human conjunctival epithelial autologous cultivated ex vivo for reconstruction of the ocular surface with symblepharon.

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of human conjunctival epithelial autologous cultivated ex vivo for reconstruction of the ocular surface in patients with symblepharon.

DETAILED DESCRIPTION:
10 patients will be included from 16 to 90 years with presence of symblepharon, what have been already subjected to proceedings of reconstruction of the ocular surface without success and to present conjunctival healthy. In the place of biopsy and after the surgery of the patient one will be applied ointment with antibiotic and corticoid to minimize the inflammatory effects. The fragments will be transported even it laboratory of Molecular Biology of the advanced Centre of Ocular Surface where it will be prosecuted by means of technique sterile under laminating flow. The conjunctival epithelias cells will be put on the amniotic membrane compartments of the plate of culture where the appropriate ways will be added. After 2 weeks the membranes colonized with epithelium conjunctival they will be subjected to the coloration and the cloth will be used for the surgery of reconstruction of the ocular surface. It will be carried out first us an evaluation ophthalmologic complete weekly, 2 months and then fortnightly up to the sixth month post-operative.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ocular surface disorders, e.g. symblepharon
* Indications for surgery will be the presence of ocular surface symptoms in the affected eye, loss of visual acuity from visual axis obscuration or irregular astigmatism, or cosmesis.
* Only one eye of a patient will be eligible for study entry.
* Patients who are adult males and females who are aged 16 or older, and are considered mentally sound
* Patients who are willing to undergo long-term follow-up, as outlined in this protocol
* Patients who have signed an informed consent form that has been approved by the SNEC Ethics Committee.

Exclusion Criteria:

* Patients less than 16 years of age
* Patients who are incapable, either by law or of mental state, of giving consent in their own right
* Patients who are either unable or unwilling to keep scheduled appointments and adhere to the other aspects of the protocol
* Patients who are pregnant or breastfeeding
* Patients with a history of drug allergy
* Patients who have received an investigational drug within 28 days preceding surgery
* Patients with intraocular pressure over 21 mmHg or history of ocular hypertension or glaucoma
* Patients who are documented to be steroid responders

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-11; Primary Completion 2008-11 (Actual); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Reconstruction of Ocular surface in patients with symblepharon | 6 months

SECONDARY OUTCOMES:
Re - reconstruction of Ocular surface in patients with symblepharon | 6 months